CLINICAL TRIAL: NCT01125072
Title: Use of Echocardiography in the Evaluation of Chest Pain in the Emergency Department
Status: Withdrawn | Type: Observational
Why Stopped: PI no longer with institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 05-264
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Chest Pain
Keywords: chest pain; echocardiography; strain imaging
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- entire cohort: patients presenting to the emergency department with chest pain and being admitted to rule out acute coronary syndrome
  Interventions: Other: Echocardiography with strain analysis

INTERVENTIONS:
Other: Echocardiography with strain analysis — Clinical routine echocardiogram with additional off line strain analysis

SUMMARY:
Chest pain is one of the most common complaints that brings a patient to the emergency department (ED). The differential diagnosis of chest pain is broad and includes cardiac as well as non-cardiac diseases. One of the initial goals in the ED evaluation of a patient presenting with chest pain is to rapidly and accurately diagnose the presence or absence of acute coronary syndrome. The diagnostic accuracy of the initial routine evaluation is often limited and results in frequent admissions for patients presenting with chest pain for further diagnostic testing.

Echocardiography has a high sensitivity and specificity for the diagnosis of acute myocardial infarction. Tissue Doppler imaging with strain and strain rate (SR) measurement is a new echocardiographic technique, which enables accurate assessment of regional left ventricular systolic and diastolic function. Prior studies have shown that abnormal strain and SR are highly sensitive markers of ischemia. Acute ischemia induces early systolic thinning and a delay in the onset of systolic thickening, a progressive decrease in the rate and degree of maximal systolic thickening, and an abnormal ischemia-related thickening which occurs after aortic valve closure. A major obstacle to the routine use of echocardiography in the ED is the need for portable studies, using heavy, bulky portable echo machines. There are currently available portable hand-held echo machines (GE-Vivid I) that produce high quality images and offer an opportunity to incorporate echocardiography into routine practice in the ED.

This study will use of early, portable echocardiography, with detailed assessment of wall motion and left ventricular function by strain and strain rate measurements, for the evaluation of chest pain in the ED. It is hypothesized that an early with detailed left ventricular function assessment will be highly sensitive and specific for the diagnosis of myocardial ischemia, and will enable rapid triage of patients who present to the ED with chest pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Chief complaint on presentation to ED: chest pain
3. Differential diagnosis includes acute coronary syndrome as determined by the Emergency physician or admitting attending.
4. Admission to the hospital required for further cardiac work up.

Exclusion Criteria:

1. Obvious noncardiac cause of the chest pain
2. Patient requires urgent intervention before echo can be obtained
3. Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the emergency department with chest pain and are admitted to rule out acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gila Perk, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU School of Medicine, Langone Medical Center, New York, New York, United States